CLINICAL TRIAL: NCT06170892
Title: Kangaroo Position in Preterm Newborn Infants Under Oxygen Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, Principal investigator, Universidade Metodista de Piracicaba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5.983.115
Record Dates: First submitted 2023-12-03; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Newborn Morbidity
MeSH Terms: interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Intervention Model Description: The newborns were placed in the kangaroo position in a single session, and the variables were identified before, during and after the application of the technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kangaroo method (Experimental): The newborns were placed in the kangaroo position in a single session, and the variables were identified before, during and after the application of the technique.
  Interventions: Other: Kangaroo method

INTERVENTIONS:
Other: Kangaroo method — The newborns were placed in the kangaroo position in a single session, and the variables were identified before, during and after the application of the technique.

SUMMARY:
The kangaroo position, which is part of the Kangaroo Method strategy, is widely used in the Neonatal Intensive Care Unit and Neonatal Intermediate Care Units and aims to promote emotional bonding, cardiorespiratory, physiological and body temperature stability, in However, there is still little scientific evidence when it comes to newborns undergoing oxygen therapy. Identify, quantify and analyze the influence of the kangaroo position on the vital signs and respiratory comfort of preterm newborns using supplemental oxygen. To collect data, a physiotherapeutic assessment form suitable for clinical analysis was used. The newborns were placed in the kangaroo position in a single session, and the variables were identified before, during and after the application of the technique.

DETAILED DESCRIPTION:
Due to the high rates of preterm newborns (PTNBs) admitted to the Neonatal Intensive Care Unit (NICU) requiring differentiated support, the Kangaroo Mother Care (MC) emerged with the intention of reducing neonatal morbidity and mortality and hospital costs. , leading to more humanized support.

MC was integrated into Humanized Care for low birth weight newborns, alleviating pain symptoms, improving the sleep-wake state, stimulating neuropsychomotor and sensory development, in addition to reducing stress.

Consisting of three stages, the first stage begins with the detection of a high-risk pregnancy until the birth of the child, and when necessary continues in the NICU or Conventional Neonatal Intermediate Care Unit (UCINCo) during the newborn's hospitalization period. born (NB), the second stage takes place at the Canguru Neonatal Intermediate Care Unit (UCINCa) where the person responsible, with the support of the multidisciplinary team, participates in most of the care carried out in the NB and finally the third stage, which covers the period of dehospitalization, as well as monitoring the development of the newborn and providing guidance to their family, monitoring occurs between the maternity ward where the patient was hospitalized and the Basic Health Unit (UBS).

Through a biopsychosocial intervention and based on the following pillars, the MC promotes welcoming newborns and their families, respect for individualities, promotion of skin-to-skin contact and involvement of the mother and father in the care of the newborn, promoting the encouraging breastfeeding and sensorimotor development, integrating the line of care for PTNBs and/or those with low birth weight (LBW), as well as their families. The kangaroo position (CP), which is part of the MC strategy, favors emotional bonding, cardiorespiratory, physiological and body temperature stability.

Newborns who need to remain hospitalized in the NICU or UCINCo may require oxygen therapy support, due to the possibility of presenting hypoxia, hyaline membrane disease, bronchopulmonary dysplasia, heart failure and pulmonary hypertension, among others.

It is extremely important to observe newborns who are using oxygen therapy, facilitating their weaning as early as possible, since, in high quantities and prolonged use, it can result in hyperoxia, especially in premature newborns, increasing risks of oxygen toxicity, reabsorption atelectasis, ventilation depression and retinopathy of prematurity13,15,16. From this perspective, this study aims to highlight the effects of the kangaroo position on the vital signs and respiratory comfort of premature and low birth weight newborns using oxygen therapy admitted to a Conventional Intermediate Neonatal Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* newborns with a gestational age of 28 to 36 weeks and 6 days,
* up to twenty-eight days of life;
* using supplemental circulating oxygen

Exclusion Criteria:

* neuromuscular disease;
* intracranial hypertension;
* intracranial hemorrhage;
* congenital heart disease
* pneumothorax;
* pneumatocele;
* active bleeding;
* mechanical ventilation

Ages: 2 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate | 1 year
  heart rate assessment on the heart monitor
respiratory frequency rate | 1 year
  assessment of respiratory rate in 60 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade do Estado do Pará, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Srinath BK, Shah J, Kumar P, Shah PS. Kangaroo care by fathers and mothers: comparison of physiological and stress responses in preterm infants. J Perinatol. 2016 May;36(5):401-4. doi: 10.1038/jp.2015.196. Epub 2015 Dec 17. PMID 26674998
- [Result] Dargahiyan Z, Ghasemi F, Karami K, Valizadeh F, Mohammadi R. A comparative study of the effects of Kangaroo care by mothers and maternal grandmothers on the vital signs of hospitalized preterm newborns: a randomized controlled clinical trial study. Trials. 2023 Apr 14;24(1):275. doi: 10.1186/s13063-023-07288-y. PMID 37059994
- [Result] El-Farrash RA, Shinkar DM, Ragab DA, Salem RM, Saad WE, Farag AS, Salama DH, Sakr MF. Longer duration of kangaroo care improves neurobehavioral performance and feeding in preterm infants: a randomized controlled trial. Pediatr Res. 2020 Mar;87(4):683-688. doi: 10.1038/s41390-019-0558-6. Epub 2019 Sep 7. PMID 31493775
- [Result] Ferber SG, Makhoul IR. Neurobehavioural assessment of skin-to-skin effects on reaction to pain in preterm infants: a randomized, controlled within-subject trial. Acta Paediatr. 2008 Feb;97(2):171-6. doi: 10.1111/j.1651-2227.2007.00607.x. Epub 2008 Jan 3. PMID 18177441
- [Result] Span LC, van Dokkum NH, Ravensbergen AG, Bos AF, Jaschke AC. Combining Kangaroo Care and Live-Performed Music Therapy: Effects on Physiological Stability and Neurological Functioning in Extremely and Very Preterm Infants. Int J Environ Res Public Health. 2021 Jun 18;18(12):6580. doi: 10.3390/ijerph18126580. PMID 34207310